CLINICAL TRIAL: NCT03653559
Title: Effect on Weight and Adiposity of "Home Meals" in Women With Overweight or Obesity
Brief Title: Effect of Consuming "Home Meals" on Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma del Estado de Mexico (Other)
Responsible Party: Principal Investigator, Antonio Laguna Camacho, Full-time Professor, Universidad Autonoma del Estado de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15CI1506014
Record Dates: First submitted 2018-08-09; First posted 2018-08-31 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial. The model tests a new dietary recommendation ("home meals" condition) against a standard dietary recommendation ("healthy meals" condition)
Who Masked: Participant
Masking Description: Participants are only aware of the study condition in which they are allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Home meals" condition (Experimental): The recommendation consists of menus with examples of breakfast, lunch and dinner based on typical preparations plus a prescription of the number of portions of the food groups that provides 1200 kcal with a distribution of 50-60% carbohydrates, 15-20% protein and < 30% lipids.
  Interventions: Behavioral: Home meals
- "Healthy meals" condition (Active Comparator): The recommendation consists of the educative graphic tool "Eatwell plate" plus a prescription of the same number of portions of the food groups for a isocaloric diet with the same macronutrient distribution as the "home meals" condition.
  Interventions: Behavioral: Healthy meals

INTERVENTIONS:
Behavioral: Home meals — Adult participants with overweight or obesity are asked to consume "home meals" during 12 weeks.
  Arms: "Home meals" condition
Behavioral: Healthy meals — Adult participants with overweight or obesity are asked to consume "healthy meals" during 12 weeks.
  Arms: "Healthy meals" condition

SUMMARY:
The current epidemic of obesity relates to the transition from traditional to industrialised diets. The present project investigates the effect on body energy of recommending the consumption of traditional "home meals", which may be a useful recommendation against obesity. A randomized controlled trial design is applied assigning participants to a recommendation of consuming during 12 weeks either "home meals" or "healthy meals." Frequency of consumption of energy-dense foods and of exercise is monitored throughout the intervention; weight and body fat are measured at baseline and at four-week intervals. The hypothesis is that consuming more frequently "home meals" reduces at least as much weight and adiposity as "healthy meals".

DETAILED DESCRIPTION:
Obesity is a global health problem that requires effective intervention. In Mexico, 2 out of 3 adults are classed as overweight or obese. Weight gain from frequent consumption of energy dense food impairs the metabolism of lipids and glucose which causes the inflammatory state that underlies development of chronic illnesses such as cardiovascular disease. Mexican women with overweight or obesity consume on average 12 times per week food rich in sugar or fat. This indicates a high prevalence of unhealthy eating habits.

Such unhealthy habits are however determined by the modern environment. The raise in food availability is associated with increase in body weight at population level. Diverse studies indicate also an increase in the number of fast food outlets together with an increase in the frequency of eating out of the home. Therefore, people are exposed to abundance of unhealthy food that leads to acquire the habit of consuming them.

The informative education on "healthy" eating is a main intervention to abate obesity levels in the population. However, the prevalence of overweight and obesity is still increasing. In fact, if this trend continues, in 2025, 32 million of Mexican adults will achieve the diagnosis of obesity.

New perspectives for intervention are needed against obesity. We propose "home meals" as a novel strategy to enhance the effectivity of educative messages on "healthy" eating that generally presents food out of their cultural context. Our definition of "home meal" considers not only the physical space where foods are consumed but also a typical socially accepted preparation based on local foods. This proposal about "home meals" is partly made because the raise of obesity in the population coincides with the replacement of traditional diet by consumption of industrialised unhealthy food.

The present project develops an intervention that compares "home meals" vs. "healthy meals" with regards to their effect on weight and body fat. The aim is to test if the recommendation of eating "home meals" has a slimming effect and how it compares to that of the standard isocaloric recommendation of eating "healthy meals." The hypothesis is that because "home meals" are culturally tailored, they would be easier to practice, and so a similar weight/body fat loss to the "healthy meals" would be at least achieved.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 25 kg/m2 or above

Exclusion Criteria:

* Presence of chronic disease

Ages: 18 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in weight and body fat | Every four weeks during 12 weeks
  Amount of weight/fat gained or lost during the intervention

SECONDARY OUTCOMES:
Change in frequency of consumption of energy-dense foods or of exercise | Every four weeks during 12 weeks
  Change in number of times a week in which participants consumed energy dense foods or exercised relative to their baseline levels

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Laguna Camacho, PhD, Principal Investigator — Universidad Autónoma del Estado de Mexico
Locations (1):
- Centro de Investigación en Ciencias Médicas, Toluca, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Materials and dataset is available in the OSF platform
Time Frame: 22 August 2019
URL: https://osf.io/uk95w/